CLINICAL TRIAL: NCT06859736
Title: Survey on the Characteristics of Traditional Medicine Syndromes in Urticaria Patients At Le Van Thinh Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: Do Thanh Sang (Other)
Responsible Party: Sponsor-Investigator, Do Thanh Sang, University of Medicine and Pharmacy at Ho Chi Minh City, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Other Study IDs: 241047 - ĐHYD
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Urticaria
MeSH Terms: conditions — Urticaria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Urticaria Patients with Traditional Medicine Syndrome Classification: This cohort includes patients diagnosed with acute or chronic urticaria who will be classified based on Traditional Medicine (TM) syndromes. Patients will be assessed using TM diagnostic criteria, including syndromes such as Blood Heat generating Wind, Blood Stagnation generating Wind, and Blood Deficiency generating Dry Wind. The study aims to evaluate the prevalence of these syndromes and their correlation with itching severity measured by the Visual Analogue Scale (VAS).

SUMMARY:
This study aims to investigate the characteristics of Traditional Medicine (TM) syndromes in urticaria patients at Le Van Thinh Hospital. Urticaria is a common dermatological condition that significantly impacts patients' quality of life. However, there is limited research on TM syndrome classification in this patient group. The study will collect data on symptoms, TM syndromes, and disease severity to determine common syndromes and their associations with clinical manifestations.

The study will be conducted as a cross-sectional, observational study with an estimated 200 participants. Eligible patients are those aged 18 years or older, diagnosed with acute or chronic urticaria, and willing to participate. The primary outcomes include the prevalence of TM syndromes, itching severity measured by the Visual Analogue Scale (VAS), and the correlation between TM syndromes and itching severity.

The study is approved by the Institutional Review Board (IRB) of the University of Medicine and Pharmacy at Ho Chi Minh City and will be conducted from December 2024 to April 2025 at Le Van Thinh Hospital, Vietnam.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 15 years or older.
* Diagnosed with acute or chronic urticaria based on modern medical criteria.
* Willing to participate and provide informed consent.

Exclusion Criteria:

* Patients with other dermatological conditions that may interfere with the diagnosis of urticaria.
* Patients currently using medications that may alter symptom presentation (e.g., antihistamines, corticosteroids, immunosuppressants).
* Patients who refuse to participate in the study

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit patients diagnosed with acute or chronic urticaria at Le Van Thinh Hospital, Vietnam. The study population will include adult patients (≥15 years old) who meet the eligibility criteria. The focus of the study is to classify Traditional Medicine (TM) syndromes in urticaria patients and explore their association with disease severity. Participants will undergo TM-based diagnostic assessment to determine the prevalence of TM syndromes such as Blood Heat generating Wind, Blood Stagnation generating Wind, and Blood Deficiency generating Dry Wind
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Traditional Medicine Syndromes in Urticaria Patients | At the time of patient enrollment (Baseline assessment, within the first visit)
  The study aims to determine the prevalence of Traditional Medicine (TM) syndromes in patients diagnosed with acute or chronic urticaria. Patients will be classified based on TM diagnostic criteria, including Blood Heat generating Wind, Blood Stagnation generating Wind, and Blood Deficiency generating Dry Wind. The percentage of patients presenting with each syndrome will be calculated.

IPD SHARING:
Plan to Share IPD: Undecided